CLINICAL TRIAL: NCT03814720
Title: VRC 321: A Phase I Open-Label Clinical Trial to Evaluate Dose, Safety, Tolerability, and Immunogenicity of an Influenza H1 Stabilized Stem Ferritin Vaccine, VRCFLUNPF099-00-VP, in Healthy Adults
Brief Title: Dose, Safety, Tolerability and Immunogenicity of an Influenza H1 Stabilized Stem Ferritin Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 190032; 19-I-0032 (Other: NIH IRB)
Record Dates: First submitted 2019-01-23; First posted 2019-01-24 (Actual); Results first posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Influenza Infection
Keywords: Flu; Seasonal Allergy; Respiratory Illness; Flu Virus; Viral Infection
MeSH Terms: conditions — Influenza, Human; Rhinitis, Allergic, Seasonal; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: H1ssF_3928 (20 mcg), ages 18-40 years (Experimental): H1ssF_3928 (20 mcg) administered intramuscularly (IM) by Needle/Syringe (Day 0)
  Interventions: Biological: VRC-FLUNPF099-00-VP (H1ssF_3928)
- Group 2A: H1ssF_3928 (60 mcg), ages 18-40 years (Experimental): H1ssF_3928 (60 mcg) administered IM by Needle/Syringe (Day 0 and Week 16)
  Interventions: Biological: VRC-FLUNPF099-00-VP (H1ssF_3928)
- Group 2B: H1ssF_3928 (60 mcg), ages 41-49 years (Experimental): H1ssF_3928 (60 mcg) administered IM by Needle/Syringe (Day 0 and Week 16)
  Interventions: Biological: VRC-FLUNPF099-00-VP (H1ssF_3928)
- Group 2C: H1ssF_3928 (60 mcg), ages 50-59 years (Experimental): H1ssF_3928 (60 mcg) administered IM by Needle/Syringe (Day 0 and Week 16)
  Interventions: Biological: VRC-FLUNPF099-00-VP (H1ssF_3928)
- Group 2D: H1ssF_3928 (60 mcg), ages 60-70 years (Experimental): H1ssF_3928 (60 mcg) administered IM by Needle/Syringe (Day 0 and Week 16)
  Interventions: Biological: VRC-FLUNPF099-00-VP (H1ssF_3928)

INTERVENTIONS:
Biological: VRC-FLUNPF099-00-VP (H1ssF_3928) — The vaccine is composed of the HA stem domain from Influenza A/New Caledonia/20/1999 (H1N1) genetically fused to the ferritin protein from H. pylori. Purified H1ssF_3928 particles display eight well-formed HA trimers that antigenically resemble the native H1 stem viral spikes.

SUMMARY:
Background:

The flu is a common viral infection that can be deadly for certain people. Vaccines against flu have been developed to teach the body to prevent or fight the infection. A new vaccine may help the body to make an immune response to H1 flu, a flu strain that infects humans.

Objective:

To test the safety and effectiveness of the H1 Stabilized Stem Ferritin vaccine (VRC-FLUNPF099-00-VP).

Eligibility:

Healthy people ages 18-70 years old who got at least 1 licensed flu vaccine since January 1, 2014.

Design:

Participants received 1 or 2 vaccinations by injections (shots) in the upper arm muscle over 4 months. Participants received a thermometer and recorded their temperature and symptoms every day a diary card for 7 days after each injection. The injection site was checked for redness, swelling, or bruising.

Participants had 9-11 follow-up visits over 12-15 months. At follow-up visits, participants had blood drawn and were checked for health changes or problems. Participants who reported influenza-like illness had nose and throat swabs for evaluation of viral infection.

Some participants had apheresis. A needle was placed into a vein in both arms. Blood was removed through a needle in the vein of one arm. A machine removed the white blood cells and then the rest of the blood was returned to the participant through a needle in the other arm.

A separate consent was provided to participants for genetic testing on their samples.

DETAILED DESCRIPTION:
Study Design: This was a Phase I, open-label, dose escalation study to evaluate the dose, safety, tolerability, and immunogenicity of VRC-FLUNPF099-00-VP in two regimens. The hypotheses were that the vaccine is safe and tolerable and will elicit an immune response. The primary objective was to evaluate the safety and tolerability of the investigational vaccine in healthy adults. Secondary objectives were related to immunogenicity of the investigational vaccine and dosing regimen.

Study Products: The investigational vaccine, VRC-FLUNPF099-00-VP (H1ssF_3928), was developed by the Vaccine Research Center (VRC), National Institute of Allergy and Infectious Diseases (NIAID) and is composed of Helicobacter pylori non-heme ferritin assembled with influenza virus H1 haemagglutinin (HA) insert to form a nanoparticle displaying eight HA stabilized stem trimers from A/New Caledonia/20/1999 (H1N1) influenza. The vaccine was supplied in single-use vials at a concentration of 180 mcg/mL. H1ssF_3928 was administered intramuscularly (IM) in the deltoid muscle via needle and syringe.

Participants: Healthy adults between the ages of 18-70 years, inclusive.

Study Plan: The study evaluated the safety, tolerability and immunogenicity of 1 or 2 doses of the H1ssF_3928 vaccine in a dose-escalation design. In Group 1, five participants received a single low dose (20 mcg) of H1ssF_3928 on Day 0. For Group 1, the protocol required 1 vaccination visit, about 9 follow-up visits, and a telephone contact after vaccination.

Once the low dose was assessed as safe and well tolerated, enrollment began for Group 2A. Groups 2A, 2B, 2C, and 2D were stratified by age as shown in the vaccination schema below. In Group 2A, participants received a higher dose (60 mcg) of H1ssF_3928 on Day 0. Once this higher dose was assessed as safe and well tolerated, participants in Group 2A received a second vaccination at Week 16 and enrollment began for Groups 2B, 2C, and 2D. For Groups 2A, 2B, 2C, and 2D, the protocol required 2 vaccination visits, about 11 follow-up visits, and a telephone contact after each vaccination. Group 2A completed the product administration schedule per protocol. While most participants in Groups 2B-2D completed the second dose administration per protocol, one participant was not able to receive the second dose due to moving out of the area and 11 participants were not able to receive their second dose due to the COVID-19 pandemic.

For all groups, solicited reactogenicity was evaluated using a 7-day diary card. Assessment of vaccine safety included clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.

VRC 321 Vaccination Schema:

Group: 1; Age Cohort: 18-40; Participants: 5; Day 0: 20 mcg

Group: 2A; Age Cohort: 18-40; Participants: 12; Day 0: 60 mcg; Week 16: 60 mcg

Group: 2B; Age Cohort: 41-49; Participants: 12; Day 0: 60 mcg; Week 16: 60 mcg

Group: 2C; Age Cohort: 50-59; Participants: 12; Day 0: 60 mcg; Week 16: 60 mcg

Group: 2D; Age Cohort: 60-70; Participants: 11*; Day 0: 60 mcg; Week 16: 60 mcg

Total: 52*

*Recruitment for the final open group, Group 2D, was ongoing to meet the accrual target of 53 participants. However, due to the COVID-19 pandemic, enrollment was discontinued with a total of 52 participants enrolled.

Study Duration:

Group 1: Participants were evaluated for 52 weeks following the vaccine administration and through an influenza season.

Groups 2A, 2B, 2C, 2D: Participants were evaluated for 52 weeks following the last vaccine administration and through an influenza season.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Healthy adults between the ages of 18-70 years inclusive
2. Based on history and examination, in good general health and without history of any of the conditions listed in the exclusion criteria
3. Received at least one licensed influenza vaccine from 2014 to the present
4. Able and willing to complete the informed consent process
5. If enrolled in Group 1: Available for clinic visits for 52 weeks after enrollment and through an influenza season
6. If enrolled in Group 2A, 2B, 2C, or 2D: Available for clinic visits for 68 weeks after enrollment and through an influenza season
7. Willing to have blood samples collected, stored indefinitely, and used for research purposes
8. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
9. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) less than or equal to 40 within the 28 days before enrollment

   Laboratory Criteria within 28 days before enrollment
10. White blood cells (WBC) and differential either within institutional normal range or accompanied by the site Principal Investigator (PI) or designee approval
11. Total lymphocyte count greater than or equal to 800 cells/mm^3
12. Platelets = 125,000 - 500,000/mm3
13. Hemoglobin within institutional normal range
14. Serum iron either within institutional normal range or accompanied by the site PI or designee approval
15. Serum ferritin within institutional normal range or accompanied by the site PI or designee approval
16. Alanine aminotransferase (ALT) less than or equal to 1.25 x institutional upper limit of normal (ULN)
17. Aspartate aminotransferase (AST) less than or equal to 1.25 x institutional ULN
18. Alkaline phosphatase (ALP) <1.1 x institutional ULN
19. Total bilirubin within institutional normal range
20. Serum creatinine less than or equal to 1.1 x institutional ULN
21. Negative for HIV infection by an FDA-approved method of detection

    Criteria applicable to women of childbearing potential:
22. Negative beta-human chorionic gonadotropin (beta-HCG) pregnancy test (urine or serum) on the day of enrollment
23. Agreed to use an effective means of birth control from at least 21 days prior to enrollment through the end of the study

EXCLUSION CRITERIA:

1. Breast-feeding or planning to become pregnant during the study.

   Participant has received any of the following substances:
2. More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment
3. Blood products within 16 weeks prior to enrollment
4. Live attenuated vaccines within 4 weeks prior to enrollment
5. Inactivated vaccines within 2 weeks prior to enrollment
6. Investigational research agents within 4 weeks prior to enrollment or planned to receive investigational products while on the study
7. Current allergy treatment with allergen immunotherapy with antigen injections, unless on maintenance schedule
8. Current anti-TB (tuberculosis) prophylaxis or therapy
9. Previous investigational H1 influenza vaccine
10. Previous investigational ferritin-based vaccine
11. Receipt of a licensed influenza vaccine within 6 weeks before trial enrollment

    Participant has a history of any of the following clinically significant conditions:
12. Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator
13. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
14. Asthma that is not well controlled
15. Diabetes mellitus (type I or II), with the exception of gestational diabetes
16. Thyroid disease that is not well controlled
17. Idiopathic urticaria within the past year
18. Autoimmune disease or immunodeficiency
19. Hypertension that is not well controlled (baseline systolic > 140 mmHg or diastolic > 90 mmHg)
20. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
21. Malignancy that is active or history of malignancy that is likely to recur during the period of the study.
22. Seizure disorder other than 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years
23. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
24. Guillain-Barré Syndrome
25. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a participant's ability to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia T Widge, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krammer F, Palese P, Steel J. Advances in universal influenza virus vaccine design and antibody mediated therapies based on conserved regions of the hemagglutinin. Curr Top Microbiol Immunol. 2015;386:301-21. doi: 10.1007/82_2014_408. PMID 25007847
- [Background] Kanekiyo M, Wei CJ, Yassine HM, McTamney PM, Boyington JC, Whittle JR, Rao SS, Kong WP, Wang L, Nabel GJ. Self-assembling influenza nanoparticle vaccines elicit broadly neutralizing H1N1 antibodies. Nature. 2013 Jul 4;499(7456):102-6. doi: 10.1038/nature12202. Epub 2013 May 22. PMID 23698367
- [Background] Yassine HM, Boyington JC, McTamney PM, Wei CJ, Kanekiyo M, Kong WP, Gallagher JR, Wang L, Zhang Y, Joyce MG, Lingwood D, Moin SM, Andersen H, Okuno Y, Rao SS, Harris AK, Kwong PD, Mascola JR, Nabel GJ, Graham BS. Hemagglutinin-stem nanoparticles generate heterosubtypic influenza protection. Nat Med. 2015 Sep;21(9):1065-70. doi: 10.1038/nm.3927. Epub 2015 Aug 24. PMID 26301691
- [Derived] Widge AT, Hofstetter AR, Houser KV, Awan SF, Chen GL, Burgos Florez MC, Berkowitz NM, Mendoza F, Hendel CS, Holman LA, Gordon IJ, Apte P, Liang CJ, Gaudinski MR, Coates EE, Strom L, Wycuff D, Vazquez S, Stein JA, Gall JG, Adams WC, Carlton K, Gillespie RA, Creanga A, Crank MC, Andrews SF, Castro M, Serebryannyy LA, Narpala SR, Hatcher C, Lin BC, O'Connell S, Freyn AW, Rosado VC, Nachbagauer R, Palese P, Kanekiyo M, McDermott AB, Koup RA, Dropulic LK, Graham BS, Mascola JR, Ledgerwood JE; VRC 321 study team. An influenza hemagglutinin stem nanoparticle vaccine induces cross-group 1 neutralizing antibodies in healthy adults. Sci Transl Med. 2023 Apr 19;15(692):eade4790. doi: 10.1126/scitranslmed.ade4790. Epub 2023 Apr 19. PMID 37075129
- [Derived] Andrews SF, Cominsky LY, Shimberg GD, Gillespie RA, Gorman J, Raab JE, Brand J, Creanga A, Gajjala SR, Narpala S, Cheung CSF, Harris DR, Zhou T, Gordon I, Holman L, Mendoza F, Houser KV, Chen GL, Mascola JR, Graham BS, Kwong PD, Widge A, Dropulic LK, Ledgerwood JE, Kanekiyo M, McDermott AB. An influenza H1 hemagglutinin stem-only immunogen elicits a broadly cross-reactive B cell response in humans. Sci Transl Med. 2023 Apr 19;15(692):eade4976. doi: 10.1126/scitranslmed.ade4976. Epub 2023 Apr 19. PMID 37075126
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-I-0032.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited at the NIH Clinical Center in Bethesda, Maryland.
Period: Overall Study
Arm/Group | Group 1: H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 Years
Started | 5 | 12 | 12 | 12 | 11
Received First Product Administration | 5 | 12 | 12 | 12 | 11
Received All Product Administrations | 5 | 12 | 7 (One participant did not receive the second dose due to moving out of area and 4 participants did not receive the second dose due to the COVID-19 pandemic) | 9 (Three (3) participants did not receive the second dose due to the COVID-19 pandemic) | 7 (Four (4) participants did not receive the second dose due to the COVID-19 pandemic)
Completed | 5 | 11 | 12 | 12 | 11
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 Years | Total
Number analyzed (Participants) | 5 | 12 | 12 | 12 | 11 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (5.6) | 29.2 (5.2) | 45.3 (3.6) | 52.8 (2.7) | 63.0 (2.5) | 46.0 (13.0)
Age, Customized [Count of Participants; unit: Participants]
  21-30 years | 2 | 8 | 0 | 0 | 0 | 10
  31-40 years | 3 | 4 | 0 | 0 | 0 | 7
  41-50 years | 0 | 0 | 12 | 3 | 0 | 15
  51-60 years | 0 | 0 | 0 | 9 | 1 | 10
  61-70 years | 0 | 0 | 0 | 0 | 10 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 7 | 7 | 6 | 28
  Male | 1 | 8 | 5 | 5 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 1 | 0 | 5
  Not Hispanic or Latino | 4 | 9 | 12 | 11 | 11 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 3 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2 | 1 | 5
  White | 4 | 8 | 7 | 10 | 10 | 39
  More than one race | 1 | 2 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.8 (2.9) | 27.0 (3.5) | 27.0 (3.7) | 27.6 (3.0) | 26.3 (4.3) | 26.6 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Each H1ssF_3928 Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, modified from FDA Guidance - September 2007.
Time Frame: 7 days after each H1ssF_3928 product administration, at approximately Week 1 and at approximately Week 17
Population: Population included all enrolled participants who received at least one H1ssF_3928 study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=52).
Measure: Count of Participants; unit: Participants
Groups:
- Overall Incidence H1ssF_3928 (20 mcg and 60 mcg): H1ssF_3928 dose groups included adults who received at least one dose of H1ssF_3928.
Arm/Group | Group 1: H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 Years | Overall Incidence H1ssF_3928 (20 mcg and 60 mcg)
Number analyzed (Participants) | 5 | 12 | 12 | 12 | 11 | 52
Participants
  Pain/Tenderness: None | 5 | 8 | 11 | 9 | 9 | 42
  Pain/Tenderness: Mild | 0 | 4 | 1 | 3 | 2 | 10
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: None | 5 | 12 | 12 | 12 | 11 | 52
  Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Redness: None | 5 | 12 | 12 | 12 | 11 | 52
  Redness: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Skin Lesion: None | 5 | 12 | 12 | 12 | 11 | 52
  Skin Lesion: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Skin Lesion: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Skin Lesion: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 5 | 8 | 11 | 9 | 9 | 42
  Any Local Symptom: Mild | 0 | 4 | 1 | 3 | 2 | 10
  Any Local Symptom: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Each H1ssF_3928 Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, modified from FDA Guidance - September 2007.
Time Frame: 7 days after each H1ssF_3928 product administration, at approximately Week 1 and at approximately Week 17
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 Years | Overall Incidence H1ssF_3928 (20 mcg and 60 mcg)
Number analyzed (Participants) | 5 | 12 | 12 | 12 | 11 | 52
Participants
  Malaise: None | 5 | 11 | 11 | 10 | 9 | 46
  Malaise: Mild | 0 | 1 | 1 | 2 | 2 | 6
  Malaise: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 4 | 10 | 12 | 11 | 11 | 48
  Myalgia: Mild | 1 | 2 | 0 | 1 | 0 | 4
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 5 | 10 | 9 | 9 | 9 | 42
  Headache: Mild | 0 | 2 | 3 | 3 | 2 | 10
  Headache: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 5 | 11 | 12 | 12 | 10 | 50
  Chills: Mild | 0 | 1 | 0 | 0 | 1 | 2
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 5 | 11 | 11 | 12 | 11 | 50
  Nausea: Mild | 0 | 1 | 1 | 0 | 0 | 2
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): None | 5 | 12 | 12 | 12 | 11 | 52
  Temperature (Fever): Mild | 0 | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): Severe | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: None | 5 | 12 | 12 | 12 | 11 | 52
  Joint Pain: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 4 | 9 | 8 | 9 | 8 | 38
  Any Systemic Symptom: Mild | 1 | 3 | 4 | 3 | 3 | 14
  Any Systemic Symptom: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following H1ssF_3928 Product Administration
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of the first study product administration through the visit scheduled for 4 weeks after each study product administration. At other time periods between study product administrations and when greater than 4 weeks after the last study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module), influenza-like illness (ILI) or influenza and new chronic medical conditions that required ongoing medical management (reported as separate outcomes) were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 4 weeks after each H1ssF_3928 product administration, up to Week 20
Population: Population included all enrolled participants who received at least one H1ssF_3928 study injection (N=52).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 Years | Overall Incidence H1ssF_3928 (20 mcg and 60 mcg)
Number analyzed (Participants) | 5 | 12 | 12 | 12 | 11 | 52
Participants
  Related to Study Product | 0 | 1 | 0 | 1 | 0 | 2
  Unrelated to Study Product | 1 | 5 | 6 | 4 | 4 | 20
  Total Number of Participants who had One or More Non-Serious Unsolicited AE | 1 | 6 | 6 | 5 | 4 | 22

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following H1ssF_3928 Product Administration
Description: SAEs were recorded from receipt of first study product administration through the last expected study visit at Week 68. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through the study participation, up to Week 68
Population: Population included all enrolled participants who received at least one H1ssF_3928 study injection (N=52).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 Years | Overall Incidence H1ssF_3928 (20 mcg and 60 mcg)
Number analyzed (Participants) | 5 | 12 | 12 | 12 | 11 | 52
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Influenza or Influenza-like Illness (ILIs) Following H1ssF_3928 Product Administration
Description: Influenza or influenza-like illness (ILI) were recorded in the study database from receipt of the first study product administration through the last study visit.
Time Frame: Day 0 through the study participation, up to Week 68
Population: Population included all enrolled participants who received at least one H1ssF_3928 study injection (N=52).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 Years | Overall Incidence H1ssF_3928 (20 mcg and 60 mcg)
Number analyzed (Participants) | 5 | 12 | 12 | 12 | 11 | 52
Participants | 0 | 1 | 0 | 3 | 0 | 4

6. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following H1ssF_3928 Product Administration
Description: New chronic medical conditions that required ongoing medical management were recorded from receipt of first study product administration through the last expected study visit at Week 68. The relationship between a new chronic medical condition and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through the study participation, up to Week 68
Population: Population included all enrolled participants who received at least one H1ssF_3928 study injection (N=52).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 Years | Overall Incidence H1ssF_3928 (20 mcg and 60 mcg)
Number analyzed (Participants) | 5 | 12 | 12 | 12 | 11 | 52
Participants
  Related to Study Product | 0 | 0 | 0 | 0 | 0 | 0
  Unrelated to Study Product | 0 | 1 | 0 | 0 | 1 | 2
  Total Number of Participants with New Chronic Medical Conditions | 0 | 1 | 0 | 0 | 1 | 2

7. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety Following H1ssF_3928 Product Administration
Description: Any abnormal laboratory results recorded after product administration as unsolicited adverse events (AEs) are summarized. Safety laboratory parameters included hematology (hemoglobin, hematocrit, platelets, and white blood cell (WBC), red blood cell (RBC), neutrophil, lymphocyte, monocyte, eosinophil and basophil percents/counts) and chemistry (alanine aminotransferase (ALT), alanine aspartate (AST), alkaline phosphate (ALP), creatinine and total bilirubin). Complete blood count (CBC) with differential, total bilirubin, AST, ALT, and ALP results were collected at Days 14, 28, 280, 364 and 476. Iron and serum ferritin were collected at Day 28. Creatinine results were collected at Day 14. Institutional laboratory normal ranges as well as the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials FDA Guidance, September 2007 were used.
Time Frame: Day 0 through the study participation, up to Week 68
Population: Population included all enrolled participants who had laboratory results available at any study visit post product administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 Years | Overall Incidence H1ssF_3928 (20 mcg and 60 mcg)
Number analyzed (Participants) | 5 | 12 | 12 | 12 | 11 | 52
Participants
  ALT | 1 | 1 | 0 | 0 | 2 | 4
  AST | 1 | 0 | 0 | 1 | 0 | 2
  WBC Count | 0 | 0 | 0 | 1 | 0 | 1
  Hemoglobin | 0 | 1 | 0 | 0 | 1 | 2
  Neutrophil Count | 0 | 0 | 2 | 1 | 0 | 3
  Lymphocyte Count | 0 | 1 | 0 | 0 | 0 | 1
  Number of Participants with one or more Abnormal Laboratory Results AE Related to Study Product | 0 | 1 | 0 | 1 | 0 | 2
  Number of Participants with one or more Abnormal Laboratory Results AE Unrelated to Study Product | 1 | 2 | 2 | 2 | 3 | 10
  Total Number of Participants who had Any Abnormal Laboratory Results Reported as AEs | 1 | 3 | 2 | 3 | 3 | 12

8. Secondary Outcome: Pseudoviral Neutralization Assay Geometric Mean Titer (GMT) Against Homologous A/New Caledonia/20/1999 Virus (H1N1) Following the Completion of Each Vaccination Regimen
Description: Pseudoviral neutralization antibody titers were determined against the homologous H1N1 A/New Caledonia/20/99 virus, and were summarized using geometric mean 80% inhibitory concentration (IC80).
Time Frame: Baseline to 2 weeks after 1st dose for participants who received a single injection, at Week 2 or From Baseline to 2 weeks after 1st dose and from Week 16 to 2 weeks after 2nd dose for participants who received two injections, at Weeks 2 and 18
Population: Baseline, Week 2, and Week 16 analyses included all who received at least one H1ssF_3928 study injection for which samples were available (N=52, 51, and 36 respectively). Week 18 analysis included all who received two H1ssF_3928 injections for which samples were available (N=32). Twelve (12) participants did not receive the 2nd injection: one Group 2B participant due to moving out of the area and 11 participants (4 in Group 2B, 3 in Group 2C and 4 in Group 2D) due to the COVID-19 pandemic.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 Years
Number analyzed (Participants) | 5 | 12 | 12 | 12 | 11
titer
  Week 0 (Baseline, Pre-Administration) | 618 [181 to 2111] | 536 [276 to 1038] | 212 [67 to 674] | 170 [108 to 269] | 283 [100 to 799]
  Week 2 (14 Days After First Product Administration): number analyzed (Participants) | 5 | 12 | 12 | 12 | 10
  Week 2 (14 Days After First Product Administration) | 916 [243 to 3454] | 888 [404 to 1949] | 566 [196 to 1632] | 651 [404 to 1051] | 741 [281 to 1955]
  Week 16 (Second Product Administration): number analyzed (Participants) | 0 | 12 | 8 | 9 | 7
  Week 16 (Second Product Administration) |  | 982 [500 to 1928] | 725 [413 to 1270] | 484 [232 to 1011] | 792 [228 to 2747]
  Week 18 (14 Days After Second Product Administration): number analyzed (Participants) | 0 | 11 | 6 | 8 | 7
  Week 18 (14 Days After Second Product Administration) |  | 602 [193 to 1876] | 780 [399 to 1526] | 543 [265 to 1112] | 894 [295 to 2706]

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after each study injection. Unsolicited AEs were recorded from receipt of the first study injection through the visit scheduled 4 weeks after each study injection. At other time periods between injections and when greater than 4 weeks after the last injection, only serious AEs, influenza or influenza-like illness (ILI) and new chronic medical conditions that required ongoing medical management were recorded through the last study visit.
Description: The overall Arms/Groups summarize AEs collected after each product administration separately and grouped by the study product and dose. Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Groups:
- Overall Incidence H1ssF_3928 (20 mcg), Ages 18-40 Years: H1ssF_3928 (20 mcg) dose group included adults (ages 18-40 years) who received a single 20 mcg dose of H1ssF_3928.
  Population included all enrolled subjects who received a H1ssF_3928 (20 mcg) study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=5).
- Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years: H1ssF_3928 (60 mcg) dose groups included adults (ages 18-40 years) who were randomized to receive two doses of 60 mcg H1ssF_3928 16 weeks apart.
  Population included all enrolled subjects who received at least one H1ssF_3928 (60 mcg) study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=12).
- Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years: H1ssF_3928 (60 mcg) dose groups included adults (ages 41-49 years) who were randomized to receive two doses of 60 mcg H1ssF_3928 16 weeks apart.
  Population included all enrolled subjects who received at least one H1ssF_3928 (60 mcg) study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=12).
- Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years: H1ssF_3928 (60 mcg) dose groups included adults (ages 50-59 years) who were randomized to receive two doses of 60 mcg H1ssF_3928 16 weeks apart.
  Population included all enrolled subjects who received at least one H1ssF_3928 (60 mcg) study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=12).
- Group 2D: H1ssF_3928 (60 mcg), Ages 60-70: H1ssF_3928 (60 mcg) dose groups included adults (ages 60-70 years) who were randomized to receive two doses of 60 mcg H1ssF_3928 16 weeks apart.
  Population included all enrolled subjects who received at least one H1ssF_3928 (60 mcg) study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=11).
- Overall Incidence H1ssF_3928 (60 mcg): H1ssF_3928 (60 mcg) dose groups included adults stratified by age (ages 18-40 years, ages 41-49 years, ages 50-59 years, and ages 60-70 years) who were randomized to receive two doses of 60 mcg H1ssF_3928 16 weeks apart.
  Population included all enrolled subjects who received at least one H1ssF_3928 (60 mcg) study injection and provided safety data (via diary card and/or laboratory results) following the injection (N=47).
Arm/Group | Overall Incidence H1ssF_3928 (20 mcg), Ages 18-40 Years | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 | Overall Incidence H1ssF_3928 (60 mcg)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/12 | 0/12 | 0/12 | 0/11 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/12 | 0/12 | 0/12 | 0/11 | 0/47
Other Adverse Events (participants affected / at risk) | 2/5 | 8/12 | 8/12 | 7/12 | 7/11 | 30/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Incidence H1ssF_3928 (20 mcg), Ages 18-40 Years (N=5) | Group 2A: H1ssF_3928 (60 mcg), Ages 18-40 Years (N=12) | Group 2B: H1ssF_3928 (60 mcg), Ages 41-49 Years (N=12) | Group 2C: H1ssF_3928 (60 mcg), Ages 50-59 Years (N=12) | Group 2D: H1ssF_3928 (60 mcg), Ages 60-70 (N=11) | Overall Incidence H1ssF_3928 (60 mcg) (N=47)
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 4
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 3
Administration site pain (General disorders) | 0 | 4 | 1 | 3 | 2 | 10
Malaise (General disorders) | 0 | 1 | 1 | 2 | 2 | 6
Headache (Nervous system disorders) | 0 | 2 | 3 | 3 | 2 | 10
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 — Joint Pain
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
All 52 participants received at least one study product administration. Groups 1 and 2A completed the product administration schedule per protocol. While most participants in Groups 2B-2D completed the second product administration per protocol, one participant was not able to receive the second dose due to moving out of the area and 11 participants were not able to receive their second dose because of visit interruptions due to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT03814720/Prot_SAP_ICF_000.pdf